CLINICAL TRIAL: NCT02931019
Title: The Effect of Head Position on the Intubating Condition Using Fiberoptic Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Sanghee Park, Clinical assistant professor, Chonnam National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CNUHH-2016-120; Institutional Review Board (Other: Chonnam National University Hwasun Hospital Institutional Review Board)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Intubation; Posture
Keywords: fiberoptic; intubation; posture
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- neck flexion first (Experimental): With specific head posture, intubation is done under flexible fiberoscopy guide.
  In this arm, at the position with neck flexion, fiberoscopy is pulled into the mouth and get the photo of laryngeal view. After then, neck position is changed to neck extension, And the laryngeal view is gotten in the same way.
  Interventions: Procedure: Intubation
- neck extension first (Experimental): In this arm, at the position with neck extension, fiberoscopy is pulled into the mouth and get the photo of laryngeal view. After then, neck position is changed to neck flexion, And the laryngeal view is gotten in the same way.
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation

SUMMARY:
For better view of fiberoptic intubation, the posture of neck is compared between neck flexion and extension.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 or 2
* scheduled for general anesthesia with endotracheal intubation
* decided to join this clinical study voluntarily

Exclusion Criteria:

* history of difficult intubation
* anticipated the difficult intubation: Total airway score > 6, upper lip bite test grade III, with cervical spine disease, history of head or neck surgery
* risk of aspiration

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
POGO score | a week (after get the picture)
  The percentage of glottic opening

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

REFERENCES:
- [Derived] Park S, Lee HG, Choi JI, Lee S, Jang EA, Bae HB, Rhee J, Yang HC, Jeong S. Comparison of vocal cord view between neutral and sniffing position during orotracheal intubation using fiberoptic bronchoscope: a prospective, randomized cross over study. BMC Anesthesiol. 2019 Jan 5;19(1):3. doi: 10.1186/s12871-018-0671-9. PMID 30611215